CLINICAL TRIAL: NCT06830577
Title: Efficacy of Intra-ureteric Aminophylline Instillation on Flexible Ureteroscopy Procedure: A Randomized Controlled Study
Brief Title: Intra-ureteric Aminophylline Instillation on Flexible Ureteroscopy Procedure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Younan Ramsis, Lecturer of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Intraureteric aminophylline
Record Dates: First submitted 2025-02-03; First posted 2025-02-17 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Stones, Kidney; Ureteric Injury
Keywords: Aminophylline; Ureteric access sheath; ureteric injury; Flexible Uretroscopy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Aminophylline Group: Intra-ureteric instillation of aminophylline (Experimental): a ureteric catheter 6 Fr will be used for instillation of normal saline supplemented with aminophylline 250 mg/10 mL at three points (Pelvi-ureteric junction, upper sacroiliac joint level and proximal to uretero-vesical junction by 5 cm) then wait for 5 minutes
  Interventions: Drug: Usage of Aminophylline prior to ureteric dilatation in Flexible uretroscopy
- Group B: Ureteral Dilator Group: Traditional ureteral dilators (Active Comparator): traditional ureteral dilators will be used. We will start by ureteral dilator 6 fr and gradually increase the size up to 12 Fr
  Interventions: Device: Sequential teflon dilator usage prior to ureteric access sheath placement in flexible uretroscopy
- Group C: Combination Group: Aminophylline instillation and Ureteral dilators (Other): Aminophylline will be instilled as in group (A) then followed by traditional ureteral dilatation as in group (B)
  Interventions: Drug: Usage of Aminophylline prior to ureteric dilatation in Flexible uretroscopy; Device: Sequential teflon dilator usage prior to ureteric access sheath placement in flexible uretroscopy; Other: Aminophylline instillation and Ureteral dilators together

INTERVENTIONS:
Drug: Usage of Aminophylline prior to ureteric dilatation in Flexible uretroscopy — Intraureteric aminophylline installation prior to ureteric dilatation
  Other Names: Intraureteric Aminophylline instillation prior to access sheath insertion
  Arms: Group A: Aminophylline Group: Intra-ureteric instillation of aminophylline; Group C: Combination Group: Aminophylline instillation and Ureteral dilators
Device: Sequential teflon dilator usage prior to ureteric access sheath placement in flexible uretroscopy — traditional ureteral dilators will be used. We will start by ureteral dilator 6 fr and gradually increase the size up to 12 Fr
  Other Names: ureteric teflon dilators prior to access sheath insertion
  Arms: Group B: Ureteral Dilator Group: Traditional ureteral dilators; Group C: Combination Group: Aminophylline instillation and Ureteral dilators
Other: Aminophylline instillation and Ureteral dilators together — Aminophylline will be instilled as in group (A) then followed by traditional ureteral dilatation as in group (B) prior to placing the ureteric access sheath
  Other Names: combination of aminophylline instillation and ureteric teflon dilators prior to access sheath insertion
  Arms: Group C: Combination Group: Aminophylline instillation and Ureteral dilators

SUMMARY:
in this study we are going to evaluate the efficacy of intra-ureteric aminophylline instillation in facilitating ureteric access sheath placement prior to flexible ureteroscopy in reducing ureteric injury rates.

DETAILED DESCRIPTION:
Urolithiasis (kidney and ureteral stones) is a common urologic condition with increasing prevalence. Flexible ureteroscopy (FURS) is a minimally invasive technique widely used for upper ureteric and renal stones. Aminophylline, a methylxanthine derivative, has been shown to relax smooth muscles and was previously used intravesically to facilitate rigid ureteroscopy with reduced complications. This study aims to assess whether intra-ureteric aminophylline instillation improves the ease of ureteral access sheath (UAS) placement during FURS and reduces ureteric injuries.

patients will be divided into 3 groups:

1. Group A (Aminophylline Group): Intra-ureteric instillation of aminophylline
2. Group B (Ureteral Dilator Group): Traditional ureteral dilators
3. Group C (Combination Group): Aminophylline instillation + Ureteral dilators follow up of the patients will be through the success rate or failure of ureteric access sheath placement, operative time, bleeding, intra/postoperative complications and stone clearance (3-week follow-up with CT scan)

ELIGIBILITY:
Inclusion Criteria:

* Upper ureteric stones or renal stones < 2 cm

Exclusion Criteria:

1. Ureteric strictures.
2. anatomic renal disorders
3. functional renal disorders
4. Urinary tract infection.
5. Coagulopathy and uncorrected bleeding disorders.
6. Prior DJ stenting
7. any contraindication for aminophylline use: (hypersensitivity to theophylline, ethylenediamine, or any component of the drug formulation, pregnancy or lactation, active peptic ulcer, presence of cardiologic diseases, presence of neurologic diseases, presence of renal impairment and presence of hepatic dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The successful placement of ureteric access sheath | intraoperative application of the access sheath
  we will assess the successful placement of ureteric access sheath in patients (that the access sheath is passed on the guide wire till the pelviureteric junction portion of the ureter after the usage of intraureteric aminophylline or teflon dilators or the usage of both.

SECONDARY OUTCOMES:
successful stone clearance | 3 weeks postoperative follow up with urinary tract multislice CT
  the stone free rate following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Younan Samir, PhD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shabayek M, Osman T, Wahb M, Elmoazen M, Osman D, Saafan A. Intravesical aminophylline instillation as an alternative for balloon dilatation prior to semi-rigid ureteroscopic management of distal ureteral stones. World J Urol. 2022 Jul;40(7):1805-1811. doi: 10.1007/s00345-022-04039-7. Epub 2022 May 26. PMID 35618855